CLINICAL TRIAL: NCT07249788
Title: Clinical Evaluation of Safety and Efficacy of Resmiterom in Patients With MASH (Metabolic Dysfunction-Associated Steato-Hepatitis) A Prospective, Open-label, Interventional Study
Brief Title: Resmiterom Efficacy & Safety in Patients With MASH
Acronym: REZMASH
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nabiqasim Industries (Pvt) Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NQ/HT/REZ/CT-003
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: MASH - Metabolic Dysfunction-Associated Steatohepatitis
Keywords: Resmetirom; MASH; Safety; Efficacy
MeSH Terms: interventions — resmetirom

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MASH targeted therapy (Experimental): MASH fibrosis stage 2 or 3
  Interventions: Drug: Resmetirom

INTERVENTIONS:
Drug: Resmetirom — 1st FDA approved MASH therapy

SUMMARY:
Phase 4 clinical trial study aims to further evaluate the safety and therapeutic efficacy of Resmetirom in Pakistani patients with fibroscan proven MASH.

ELIGIBILITY:
Inclusion Criteria:

* • At least one metabolic comorbidity (e.g., T2DM, obesity, dyslipidemia and hypertension)

  * Clinical diagnosis of MASH using:

    * LSM ≥ 8.5kpa And/or
    * FAST score ≥0.67 And/or
    * FibroScan CAP ≥ 275 dB/m And/or
    * FIB-4 > 1.3

Exclusion Criteria:

* • History of drug addiction and alcoholism

  * Cirrhosis or decompensated liver disease
  * Chronic viral hepatitis HBV, HCV)
  * MACE including MI, Stroke, PE etc.
  * Pregnant/lactating women
  * Concurrent use of other investigational drugs
  * History of other liver diseases (viral, autoimmune, drug-induced, alcohol)
  * Previous use of resmetirom in last 6 months
  * Significant renal impairment (eGFR <30)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2025-10-17 (Actual); Primary Completion 2026-10-16 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
FIB-4 and CAP score/LSM on fibroscan | 6 months
  Changes in liver fibrosis using non invasive markers
Changes in thyroid profile | 6 months
  thyroid profile of each patient at baseline and at primary end point

CONTACTS AND LOCATIONS:
Locations (1):
- Liver transplant center, Holy family hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
Its undecided for now will be updated laterwards

REFERENCES:
- [Background] Patel RH, Parikh C, Upadhyay H, Sonaiya S, Ramnath P, Singh S, Patel U, Kothari T. Resmetirom in the Management of Metabolic Dysfunction-Associated Steatohepatitis (MASH): A Comprehensive Review of Current Evidence and Therapeutic Potential. Cureus. 2024 Nov 29;16(11):e74772. doi: 10.7759/cureus.74772. eCollection 2024 Nov. PMID 39735033
- [Background] Younossi ZM, Stepanova M, Taub RA, Barbone JM, Harrison SA. Hepatic Fat Reduction Due to Resmetirom in Patients With Nonalcoholic Steatohepatitis Is Associated With Improvement of Quality of Life. Clin Gastroenterol Hepatol. 2022 Jun;20(6):1354-1361.e7. doi: 10.1016/j.cgh.2021.07.039. Epub 2021 Jul 27. PMID 34329774
- [Background] Harrison SA, Bashir MR, Guy CD, Zhou R, Moylan CA, Frias JP, Alkhouri N, Bansal MB, Baum S, Neuschwander-Tetri BA, Taub R, Moussa SE. Resmetirom (MGL-3196) for the treatment of non-alcoholic steatohepatitis: a multicentre, randomised, double-blind, placebo-controlled, phase 2 trial. Lancet. 2019 Nov 30;394(10213):2012-2024. doi: 10.1016/S0140-6736(19)32517-6. Epub 2019 Nov 11. PMID 31727409
- [Result] Harrison SA, Bedossa P, Guy CD, Schattenberg JM, Loomba R, Taub R, Labriola D, Moussa SE, Neff GW, Rinella ME, Anstee QM, Abdelmalek MF, Younossi Z, Baum SJ, Francque S, Charlton MR, Newsome PN, Lanthier N, Schiefke I, Mangia A, Pericas JM, Patil R, Sanyal AJ, Noureddin M, Bansal MB, Alkhouri N, Castera L, Rudraraju M, Ratziu V; MAESTRO-NASH Investigators. A Phase 3, Randomized, Controlled Trial of Resmetirom in NASH with Liver Fibrosis. N Engl J Med. 2024 Feb 8;390(6):497-509. doi: 10.1056/NEJMoa2309000. PMID 38324483
- See also: Related Info — https://www.nabiqasim.com/wp-content/uploads/2025/05/Rezna-Tablets-Leaflet-Rev-03-25-0.pdf